CLINICAL TRIAL: NCT02951104
Title: Noninvasive Cardiac Output Monitoring in Pulmonary Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Santa Barbara Cottage Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-61
Record Dates: First submitted 2016-10-27; First posted 2016-11-01 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Drug Delivery Systems

ARMS (1):
- USCOM (Experimental)
  Interventions: Device: Ultrasonic Cardiac Output Monitor (USCOM) system

INTERVENTIONS:
Device: Ultrasonic Cardiac Output Monitor (USCOM) system

SUMMARY:
Comparison of Ultrasonic Cardiac Output Monitor (USCOM) system with Fick and thermodilution methods during right heart catheterization in patients with pulmonary hypertension.

ELIGIBILITY:
Inclusion criteria:

* Age > 18 years
* Diagnosis of Group 1 or Group 4 PAH based on PAPm > 25 mmHg, PAWP <15 mmHg, PVR >3 WU and consistent clinical history. Note: for logistical reasons, patients at high suspicion for Group 1 or Group 4 PAH will sign informed consent to have the USCOM system applied during right heart catheterization before the procedure; if it is found that the patient does not meet the definition of Group 1 or Group 4 PAH during right heart catheterization, he/she will be excluded.
* Willingness and ability to comply with study procedures.
* No known hypersensitivity to the components of USCOM electrodes

Exclusion criteria:

* Unwillingness to sign informed consent or inability or unwillingness to comply with study procedures
* Evidence of postcapillary pulmonary hypertension on right heart catheterization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Cardiac output measurement correlation at baseline | 30 minutes
  Correlation between cardiac output measurement between USCOM system and Fick and thermodilution methods of cardiac output measurement (standard of care)

SECONDARY OUTCOMES:
Cardiac output measurement correlation after vasodilator testing | 30 minutes
  Correlation between cardiac output measurement between USCOM system and Fick and thermodilution methods of cardiac output measurement (standard of care) after vasodilator trial testing

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Barbara Cottage Hospital, Santa Barbara, California, United States